CLINICAL TRIAL: NCT02072551
Title: Devenir au Long Cours de la Cellule bêta Chez Les Adultes Porteurs d'Anomalies génétiques à l'Origine du Diabète Néonatal
Brief Title: Future of Beta Cells in Adults With Genetic Abnormality Behind Neonatal Diabetes
Acronym: GLUCONEO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: GLUCONEO
Record Dates: First submitted 2013-11-04; First posted 2014-02-26 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- Adult with neonatal diabetes: Adult with neonatal diabetes (before 1 year ) and need for insulin
- non diabetic adults with a relative with neonatal diabetes

SUMMARY:
The main objective of this study is to evaluate Beta cells in patients with a neonotal diabetes linked to a genetic abnormality Metabolic caracteristics will described using a transversal cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18 à 65 year
* diabetic patient with a neonatal diabetis (before 1 year old) and need for insuline or patient with a relative having neonatal diabetis

Exclusion Criteria:

Diabète induit (médicaments - ex corticoïdes) ou syndromique

* infection
* cancer
* pegnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diabetic people
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Mean insulin secretion output | Week after inclusion

SECONDARY OUTCOMES:
insulin secretion outout after arginine perfusion | during hospitalisation (3 days)
sensitivity to insulin | during hospitalisation (3 days)
glucago secretion output | during hospitalisation (3 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Siant-louis, Paris, France

REFERENCES:
- [Derived] Le Bourgeois F, Beltrand J, Baz B, Julla JB, Riveline JP, Simon A, Flechtner I, Ait Djoudi M, Fauret-Amsellem AL, Vial Y, Scharfmann R, Sommet J, Boudou P, Cave H, Polak M, Gautier JF, Busiah K; TNDM Long-Term Follow-Up Study Group. Long-term Metabolic and Socioeducational Outcomes of Transient Neonatal Diabetes: A Longitudinal and Cross-sectional Study. Diabetes Care. 2020 Jun;43(6):1191-1199. doi: 10.2337/dc19-0324. Epub 2020 Apr 9. PMID 32273272